CLINICAL TRIAL: NCT02736565
Title: Phase I Trial of Pbi-shRNA™ EWS/FLI1 Type 1 Lipoplex (LPX) in Subjects With Advanced Ewing's Sarcoma
Brief Title: Pbi-shRNA™ EWS/FLI1 Type 1 LPX in Subjects With Advanced Ewing's Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gradalis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CL-PTL-001
Record Dates: First submitted 2016-04-04; First posted 2016-04-13 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Ewing's Sarcoma; Ewing Family of Tumors; Ewing's Tumor Metastatic; Ewing's Sarcoma Metastatic; Ewing's Tumor Recurrent; Rare Diseases; Sarcoma
Keywords: bone cancer; EWS gene; neuroectodermal tumor; pNET; sarcoma; soft tissue; ESFT; Immunotherapy
MeSH Terms: conditions — Sarcoma, Ewing; Neuroectodermal Tumors, Primitive, Peripheral; Rare Diseases; Sarcoma; Bone Neoplasms; Neuroectodermal Tumors; Neuroectodermal Tumors, Primitive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort -1 (Experimental): 0.02mg/kg pbi-shRNA™ EWS/FL/I1 Type 1 Lipoplex
  Interventions: Biological: pbi-shRNA™ EWS/FLI1 Type 1 Lipoplex
- Cohort 0 (Experimental): 0.03mg/kg pbi-shRNA™ EWS/FL/I1 Type 1 Lipoplex
  Interventions: Biological: pbi-shRNA™ EWS/FLI1 Type 1 Lipoplex
- Cohort 1 (Experimental): 0.04mg/kg pbi-shRNA™ EWS/FL/I1 Type 1 Lipoplex
  Interventions: Biological: pbi-shRNA™ EWS/FLI1 Type 1 Lipoplex
- Cohort 2 (Experimental): 0.06mg/kg pbi-shRNA™ EWS/FL/I1 Type 1 Lipoplex
  Interventions: Biological: pbi-shRNA™ EWS/FLI1 Type 1 Lipoplex
- Cohort 3 (Experimental): 0.08mg/kg pbi-shRNA™ EWS/FL/I1 Type 1 Lipoplex
  Interventions: Biological: pbi-shRNA™ EWS/FLI1 Type 1 Lipoplex
- Cohort 4 (Experimental): 0.10mg/kg pbi-shRNA™ EWS/FL/I1 Type 1 Lipoplex
  Interventions: Biological: pbi-shRNA™ EWS/FLI1 Type 1 Lipoplex
- Cohort 5 (Experimental): 0.125mg/kg pbi-shRNA™ EWS/FL/I1 Type 1 Lipoplex
  Interventions: Biological: pbi-shRNA™ EWS/FLI1 Type 1 Lipoplex
- Cohort 6 (Experimental): 0.156mg/kg pbi-shRNA™ EWS/FL/I1 Type 1 Lipoplex
  Interventions: Biological: pbi-shRNA™ EWS/FLI1 Type 1 Lipoplex

INTERVENTIONS:
Biological: pbi-shRNA™ EWS/FLI1 Type 1 Lipoplex — Lipoplex is given intravenously as a single administration twice a week for 4 weeks for a total of 8 infusions per cycle followed by 2 weeks of rest. Treatment may continue as long as there is clinical benefit, no evidence of disease progression, and no other withdrawal criteria are met.
  First dose started on Cycle 1 Week 1 Day 1 followed by observation and safety assessment for 13 days. If no toxicity was observed, then another single administration of study agent was given at Cycle 1 Week 3 Day 1 followed by observation and safety for 6 days. If no toxicity was observed, then study agent was given twice a week on Days 1 and 4 over 3 weeks, for a total of 8 infusions per cycle, followed by a 2-week washout before starting each subsequent cycle. Cycle 1 = 8 weeks. Each subsequent cycles = 6 weeks.
  Other Names: Lipoplex

SUMMARY:
The purpose of this study is to determine the safety and the maximum tolerated dose of of pbi-shRNA™ EWS/FLI1 Type 1 lipoplex in patients with advanced Ewing's sarcoma.

DETAILED DESCRIPTION:
Eligible participants with advanced Ewing's sarcoma will be accrued in 3-subject dose escalation cohorts using the following escalation schema (50%→33%→25%→25%→25%) at a starting IV dose of 0.04 mg/kg and up to a dose of 0.156mg/kg.

For this first in class study of pbi-shRNA™ EWS/FLI1 Type 1 lipoplex, Dose Limiting Toxicity (DLT) will be defined as any ≥ Grade 3 toxicity reported within the four weeks following the first administration of the investigational product, regardless of attribution. Any other ≥ Grade 3 toxicity encountered after the first four weeks post Dose 1 on Cycle 1 will be reported according to the CTCAE Version 4.0 but not defined as DLTs.

If 1 of 3 subjects within a dose cohort experiences a DLT, that dose cohort will be expanded to six subjects provided no further subjects experience a DLT. If no further subjects experience a DLT, dose-escalation may continue. If ≥2 subjects within a dose cohort experiences a DLT, this will define the DLT dose level and the Maximum Tolerated Dose (MTD) will have been exceeded.

The preceding dose level will be expanded to a total of 6 subjects and, if ≤1 subject experiences a DLT, that dose level will be considered the MTD. If no further subjects experience a DLT, dose-escalation may resume per escalation schema. Once the presumptive MTD is reached, an additional 6 subjects will be treated at that dose, designated the expanded MTD dose cohort.

Participants who experience an unrelated Grade ≥3 toxicity that normalizes within 1 week may continue study treatment when the adverse event returns to Grade 1 or better at 50% of their assigned cohort dose. Delay in dosing of >24 hours will require that the next dose is skipped.

As of protocol Amendment No. 5, two subjects met the definition of dose limiting toxicity at Cohort 1, 0.04mg/kg, therefore the dose reduced by 50% and subsequent lipoplex administrations were given at 0.02mg/kg. Administration of 0.02mg/kg is defined as Cohort -1. An additional 6 subjects will be treated at Cohort -1, designated the expanded MTD dose cohort. If no further subjects experience a DLT at Cohort -1, dose re-escalation may continue to Cohort 0. The dose administered for subjects in Cohort 0 is 0.03mg/kg and would be defined as the optimal dose.

All study agent administrations will cease for the occurrence of any of the following events at any time point over the four weeks following the first study agent dose administration to a participant: death, hospitalization for reasons other than those related to the participant's malignancy (excluding preplanned hospitalization and/or hospitalization for observation during the participant's first infusion), or any Grade ≥3 liver toxicity or Grade ≥4 pulmonary toxicity. All Grade ≥3 liver toxicities or Grade ≥4 pulmonary toxicities will be considered Adverse Events of Special Interest (AESI).

Participants will receive an intravenous infusion twice a week for 4 weeks for a total of 8 infusions per cycle followed by 2 weeks of rest. Treatment with investigational product may continue as long as there is clinical benefit, no evidence of disease progression, and no other withdrawal criteria are met.

Safety assessments will include physical examinations, performance status, laboratory assessments, and vital signs. Toxicity (Adverse Events) will be recorded for the duration of the participant's study treatment (following the first dose), and for up to 60 days following the last study treatment. Toxicities and AEs will be graded and reported using the Common Toxicity Criteria for Adverse Events (CTCAE) Version 4.0.

Efficacy assessments (response and progression) will be evaluated by local investigators using the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.

ELIGIBILITY:
Subjects will be eligible for registration if they meet all of the following inclusion criteria:

Inclusion Criteria:

1. Histologically confirmed Ewing's Sarcoma Family of Tumors (ESFT).
2. Age ≥8 years.
3. Evidence of EWS translocation fusion by FISH or RT-PCR or NGS.
4. Evidence of Type 1 fusion by molecular diagnostics.
5. Refractory or intolerant to standard of care. Subjects must have failed surgery (if resectable), radiation (if no function-preserving surgical approach at primary site, unresectable primary following induction chemotherapy, residual microscopic or gross disease after surgery or inadequate margins), and the following chemotherapy agents: doxorubicin, vincristine, cyclophosphamide, ifosfamide, etoposide.
6. ECOG performance status (PS) = 0-2, or Karnofsky PS ≥60% or Lansky PS ≥60%.
7. Normal organ and marrow function as defined below:

   Absolute granulocyte count ≥1,000/mm3 Absolute lymphocyte count ≥400/mm3 Platelets ≥100,000/mm3 Total bilirubin ≤ institutional upper limit of normal AST(SGOT)/ALT(SGPT) ≤2x institutional upper limit of normal Creatinine <1.5 mg/dL
8. Normal pulmonary function as defined as FEV1/FVC greater than 70% in adults or greater than 80% in individuals between 8 and 18 years of age.
9. Subject has recovered to CTCAE Grade 1 or better from all adverse events associated with prior therapy or surgery. Pre-existing motor or sensory neurologic pathology or symptoms must be recovered to CTCAE Grade 2 or better.
10. If female of childbearing potential, has a negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a negative serum test will be required for study entry.
11. Ability to understand and the willingness to sign a written informed protocol specific consent. Pediatric patients must sign an assent with a parent or legal guardian sign a written informed consent, per institutional guidelines.

Subjects will NOT be eligible for study registration and enrollment if meeting any of the following criteria:

Exclusion Criteria:

1. Anti-cancer chemotherapy, biologic therapy or immunotherapy within 3 weeks or radiation therapy within 2 weeks of first infusion.
2. Known history of other malignancy unless having undergone curative intent therapy without evidence of that disease for ≥ 3 years except cutaneous squamous cell and basal cell skin cancer, superficial bladder cancer, in situ cervical cancer or other in situ cancers are allowed if definitively resected.
3. Patients with PET avid disease only will be excluded.
4. Brain metastases unless treated with curative intent (gamma knife or surgical resection) and without evidence of progression for ≥ 2 months.
5. History of or current evidence of thrombosis.
6. History of or current evidence of any condition (including medical, psychiatric or substance abuse disorder), therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the Investigator.
7. Known HIV or chronic Hepatitis B or C infection.
8. Have signs and symptoms consistent with an active infection.
9. Live vaccination for the prevention of infectious disease administered <30 days prior to the start of study therapy or inactivated vaccination <14 days prior to the start of study therapy.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2020-08-04 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | From first dose and up to 60 days following the last treatment, up to approximately 13 months.
  Adverse events(AEs) will be recorded for the duration of the participant's study treatment (following the first dose of the investigational product), and for up to 60 days following the last study treatment. AEs will be graded and reported using the Common Toxicity Criteria for Adverse Events (CTCAE) Version 4.03. The relationship of each event to the investigational product will be assessed by the Treating Physician.
Determine the maximum tolerated dose of intravenous administration of lipoplex | From first subject, first dose and after an additional 6 subjects have been treated at the MTD, up to 4 weeks.
  By observing the Dose Limiting Toxicities, including ≥ Grade 3 toxicity encountered within the four weeks following the first administration of the investigational product the MTD will be determined.

SECONDARY OUTCOMES:
To assess disease response for different cohorts following pbi-shRNA™ EWS/FLI1 Type 1 lipoplex administration at different dose(s). | From Baseline and quarterly thereafter until progressive disease is noted, up to approximately 12 months.
  Radiological assessment of tumors, chest, abdomen, and pelvis to include, at a minimum, CT (or MRI), used to evaluate measurable or non-measurable disease. To be obtained at baseline and quarterly thereafter (+/- 4 weeks) until progressive disease is noted. For those subjects with CT or MRI evidence of response following the administration of the study agent, a confirmatory scan will be performed one month later.
To assess the pharmacokinetics of pbi-shRNA™ EWS/FLI1 Type 1 plasmid. | From Cycle 1 Week 1 Day 1 and until Cycle 2 Week 1 Day 1, approximately 8 weeks.
  Serum for pharmacokinetics (PK) analysis will be collected on Cycle 1 Week 1 Day 1, Cycle 1 Week 6 Day 4, and Cycle 2 Week 1 Day 1 at the following time points (±10%): 30 minutes prior to study agent administration and at the following time points after the initiation of study agent administration: 5 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 24 hours and 48 hours.
To assess ctDNA (EWSR-FLI1) levels and compare to tumor burden and disease response prior to and following pbi-shRNA™ EWS/FLI1 Type 1 lipoplex administration. | From Cycle 1 Week 1 Day 1 and until the last even cycle where product was administered, up to approximately 1 year.
  Blood for circulating tumor DNA analysis will be collected at Cycle 1 Week 1 Day 1, Cycle 1 Week 3 Day 1, Cycle 2 Week 1 Day 1 prior to product infusion and every even cycle thereafter at Week 1 Day 1 prior to product infusion.

CONTACTS AND LOCATIONS:
Overall Officials: John Nemunaitis, MD, Study Director — Gradalis, Inc.
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Mary Crowley Cancer Research Centers, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barve M, Wang Z, Kumar P, Jay CM, Luo X, Bedell C, Mennel RG, Wallraven G, Brunicardi FC, Senzer N, Nemunaitis J, Rao DD. Phase 1 Trial of Bi-shRNA STMN1 BIV in Refractory Cancer. Mol Ther. 2015 Jun;23(6):1123-1130. doi: 10.1038/mt.2015.14. Epub 2015 Jan 26. PMID 25619726
- [Background] Wang Z, Rao DD, Senzer N, Nemunaitis J. RNA interference and cancer therapy. Pharm Res. 2011 Dec;28(12):2983-95. doi: 10.1007/s11095-011-0604-5. Epub 2011 Oct 19. PMID 22009588
- [Background] Senzer N, Barve M, Kuhn J, Melnyk A, Beitsch P, Lazar M, Lifshitz S, Magee M, Oh J, Mill SW, Bedell C, Higgs C, Kumar P, Yu Y, Norvell F, Phalon C, Taquet N, Rao DD, Wang Z, Jay CM, Pappen BO, Wallraven G, Brunicardi FC, Shanahan DM, Maples PB, Nemunaitis J. Phase I trial of "bi-shRNAi(furin)/GMCSF DNA/autologous tumor cell" vaccine (FANG) in advanced cancer. Mol Ther. 2012 Mar;20(3):679-86. doi: 10.1038/mt.2011.269. Epub 2011 Dec 20. PMID 22186789
- [Background] Rao DD, Jay C, Wang Z, Luo X, Kumar P, Eysenbach H, Ghisoli M, Senzer N, Nemunaitis J. Preclinical Justification of pbi-shRNA EWS/FLI1 Lipoplex (LPX) Treatment for Ewing's Sarcoma. Mol Ther. 2016 Aug;24(8):1412-22. doi: 10.1038/mt.2016.93. Epub 2016 May 11. PMID 27166877